CLINICAL TRIAL: NCT01642407
Title: A Phase 3, Multi-center, Open-label Study To Investigate Safety, Efficacy, And Tolerability Of Sildenafil Citrate In Pediatric Patients With Pulmonary Arterial Hypertension
Brief Title: Safety And Efficacy Of Sildenafil In Children With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1481298
Record Dates: First submitted 2012-06-15; First posted 2012-07-17 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension; Hypertension, Pulmonary
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sildenafil (Experimental)
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Body weight > 20 kg: 20 mg TID (60 mg/day) Body weight ≤ 20 kg: 10 mg TID (30 mg/day) Treatment duration: 16 weeks in Part 1, until until sildenafil obtained marketing approval in Part 2

SUMMARY:
Pulmonary arterial hypertension (PAH) is a rare, progressive, and life-threatening disease. In many patients, the course of PAH is a steady deterioration and reduced life expectancy.

Sildenafil was approved by the European Commission for the treatment of PAH in pediatric patients in May 2011, making it the first agent to be approved for the treatment of children with PAH. The approval was based on the largest placebo-controlled study to be conducted in this population. The recommended dose in pediatric patients aged 1 year to 17 years old is 10 mg TID in patients ≤ 20 kg and 20 mg TID for patients > 20 kg. Higher doses are not recommended in pediatrics patients.

This study is an open-label, multi-center study to investigate safety, efficacy and pharmacokinetics of sildenafil citrate in Japanese pediatric patients with PAH.

ELIGIBILITY:
Inclusion Criteria:

* Subjects weighing ≥8 kg.
* Subjects who have symptomatic pulmonary arterial hypertension due to one of the following conditions:
* Idiopathic pulmonary arterial hypertension; or
* Heritable pulmonary arterial hypertension; or
* Pulmonary arterial hypertension associated with congenital systemic-to-pulmonary shunts. If the defect(s) is repaired, the subject's condition should be stabilized hemodynamically; or
* Pulmonary arterial hypertension associated with d-transposition of the great arteries repaired within the first 30 days of life; or
* Pulmonary arterial hypertension in subjects who have undergone surgical repair of other congenital heart lesions and the condition should be stabilized hemodynamically and do not have clinically significant residual left-sided heart disease.
* Subjects with a mean pulmonary artery pressure ≥25 mmHg at rest, PCWP ≤15 mmHg, and PVRI ≥3 Wood units x m2. If PCWP is not available, then mean LA pressure ≤15 mmHg or LVEDP ≤15 mmHg in the absence of left atrial obstruction.

Exclusion Criteria:

* Left-sided heart disease.
* Subjects with Down syndrome.
* Subjects with Obstructive Sleep Apnea, regardless of treatment status.
* Pericardial constriction.
* Subjects with significant (2+ for regurgitation) valvular disease other than tricuspid or pulmonary regurgitation.
* Acutely decompensated heart failure within previous 30 days from screening.
* Subjects who have had an atrial septostomy within previous 6 months of screening.
* Subjects with hemodynamic instability or hypo- or hypertension at screening.
* Subjects with a history of stroke, myocardial infarction or life threatening arrhythmia within 6 months of screening.
* Subjects with moderate to severe restrictive pulmonary disease (Total Lung Capacity or Forced Vital Capacity ≤60% of normal) or history of severe lung disease.
* Subjects with bronchopulmonary dysplasia (BPD) and other chronic lung diseases.
* Subjects with history of pulmonary embolism.
* Subjects with known hereditary degenerative retinal disorders (such as retinitis pigmentosa) or history of non-arteritic anterior ischemic optic neuropathy (NAION).
* Subjects who are known to be HIV positive.
* Subjects with impairment of renal function (serum creatinine >2.5 × ULN) or hepatic function (ALT and/or AST >3 × ULN; and/or bilirubin ≥2 mg/dL). Hematological abnormalities (e.g., severe anemia, Hgb <10 g/dL, leukopenia, WBC <2500/µL).
* Subjects with severe hepatic dysfunction (Child-Pugh classification C).
* Change in class of medication for CHF or PAH within the 10 days prior to qualifying right heart catheterization.
* Subjects who are currently prescribed and/or taking nitrates or nitric oxide donors in any form.
* Subjects taking chronic arginine supplementation.
* Subjects who have received parenteral inotropic medication or parenteral vasodilators within 30 days of Day 1.
* Subjects who are receiving alpha-blockers, nicorandil, amiodarone or potent cytochrome P450 3A4 inhibitors.
* Subjects receiving chronic treatment with off-label sildenafil within 30 days of Day 1 are excluded. Subjects receiving an endothelin antagonist，PED5 inhibitor or, prostacyclin/prostacyclin analogue within 30 days of randomization are excluded except for beraprost.
* Pregnant females; breastfeeding females; males and females of childbearing potential not using highly effective contraception or not agreeing to continue highly effective contraception for at least 28 days after last dose of investigational product.
* Current or past illicit drug use or alcoholism excepting if abstinence can be documented for ≥1 year.
* Participation in another clinical trial of an investigational drug or device (including placebo) within 30 days of screening for entry into the present study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2012-08-24 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Japan (5):
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Osaka University Hospital, Suita, Osaka
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
  - Shizuoka Children's Hospital, Shizuoka

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481298&StudyName=Safety%20And%20Efficacy%20Of%20Sildenafil%20In%20Children%20With%20Pulmonary%20Arterial%20Hypertension

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted at 3 sites in Japan. Data reported is based on data cut-off date of 26 December 2016.
Groups:
- Sildenafil: Participants received 10 milligram (mg) or 20 mg of Sildenafil (based on their body weight) orally, thrice daily on Day 1 (Baseline), Weeks 4, 8, and 16 in Part 1 of the study. Participants who completed Part 1 and required continuing treatment with Sildenafil, received 10 mg or 20 mg of Sildenafil (based on their body weight) orally, thrice daily on Weeks 28, 40, 52 and thereafter every 12 weeks until Sildenafil obtained marketing approval (up to a maximum of 119.6 weeks). Participants with less than or equal to (<=) 20 kilogram (kg) of body weight received 10 mg dose, thrice daily as powder for oral suspension and participants with greater than (>) 20 kg of body weight received 20 mg dose, thrice daily as film-coated tablets.
Period: Part 1 (Screening Till Week 16)
Arm/Group | Sildenafil
Started | 6
Completed | 3
Not Completed | 3
Not completed — Insufficient clinical response | 3
Period: Part 2(Week17 to Maximum of 119.6 Weeks)
Arm/Group | Sildenafil
Started | 3
Completed | 1
Not Completed | 2
Not completed — Coil Embolization | 1
Not completed — Change of treatment plan | 1

BASELINE CHARACTERISTICS:
Population: Efficacy analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Sildenafil: Participants received 10 mg or 20 mg of Sildenafil (based on their body weight) orally, thrice daily on Day 1 (Baseline), Weeks 4, 8, and 16 in Part 1 of the study. Participants who completed Part 1 and required continuing treatment with Sildenafil, received 10 mg or 20 mg of Sildenafil (based on their body weight) orally, thrice daily on Weeks 28, 40, 52 and thereafter every 12 weeks until Sildenafil obtained marketing approval (up to a maximum of 119.6 weeks). Participants with <= 20 kg of body weight received 10 mg dose, thrice daily as powder for oral suspension and participants with > 20 kg of body weight received 20 mg dose, thrice daily as film-coated tablets.
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.7 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulmonary Vascular Resistance Index (PVRI) at Week 16
Description: PVRI equals pulmonary vascular resistance (PVR) times body surface area (BSA) (PVRI = PVR*BSA). PVR is the resistance to blood flow through the pulmonary circulation and it was measured in Wood units. Wood unit =80 dyne*seconds per centimetre^5 (dyne*sec/cm^5).
Time Frame: Baseline, Week 16
Population: Efficacy analysis set included all participants who received at least 1 dose of study drug. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points."
Measure: Mean (Standard Deviation); unit: wood units*meter^2
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
wood units*meter^2
  Baseline | 18.567 (11.7629)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | -4.113 (6.3770)

2. Primary Outcome: Change From Baseline in Mean Pulmonary Artery Pressure (mPAP) at Week 16
Description: It was a hemodynamic parameter and measured using a pressure transducer positioned at the mid-axillary line with the participant in the supine position.
Time Frame: Baseline, Week 16
Population: Efficacy analysis set included all participants who received at least 1 dose of study drug. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
millimeter of mercury (mmHg)
  Baseline | 58.5 (22.94)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | -6.5 (15.15)

3. Primary Outcome: Change From Baseline in World Health Organization (WHO) Functional Class in Participants With Pulmonary Arterial Hypertension (PAH) at Week 4
Description: WHO functional classification for PAH range from Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity) and Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest). The change from baseline in WHO functional class was classified into "Improved", "No change" and "Worsened". Improvement = reduction in functional class, worsened = increase in functional class and no change = no change in functional class. Change from baseline in number of participants in each functional class were reported.
Time Frame: Baseline, Week 4
Population: Efficacy analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
participants
  Baseline: Class I | 2 (0.58)
  Baseline: Class II | 3 (0.58)
  Baseline: Class III | 1
  Baseline: Class IV | 0
  Week 4: Improved | 1
  Week 4: No change | 5
  Week 4: Worsened | 0

4. Primary Outcome: Change From Baseline in World Health Organization (WHO) Functional Class in Participants With Pulmonary Arterial Hypertension (PAH) at Week 8
Description: as for outcome 3
Time Frame: Baseline, Week 8
Population: Efficacy analysis set included all participants who received at least 1 dose of study drug. Here,'N' (Overall number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 5
participants
  Improved | 1 (0.71)
  No change | 4
  Worsened | 0

5. Primary Outcome: Change From Baseline in World Health Organization (WHO) Functional Class in Participants With Pulmonary Arterial Hypertension (PAH) at Week 16
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: Efficacy analysis set included all participants who received at least 1 dose of study drug. Here, Overall Number of participants analyzed signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 4
participants
  Improved | 1 (0.71)
  No change | 3
  Worsened | 0

6. Primary Outcome: Change From Baseline in Brain Natriuretic Peptide (BNP) at Week 16
Description: BNP is produced by ventricular cardiomyocytes. It causes reduction in preload and blood pressure by vasodilatation.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picogram per milliliter
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
picogram per milliliter
  Baseline | 132.62 (135.080)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | -64.10 (129.638)

7. Primary Outcome: Change From Baseline in N-terminal Pro Brain Natriuretic Peptide (NT Pro-BNP) at Week 16
Description: NT pro-BNP is a cardiac marker, having the prognostic value for participants with heart failure or left ventricular dysfunction. Higher level of the marker was indicative of heart damage.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picogram per milliliter
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
picogram per milliliter
  Baseline | 843.03 (1120.900)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | -546.85 (1107.621)

8. Secondary Outcome: Change From Baseline in World Health Organization (WHO) Functional Class in Participants With Pulmonary Arterial Hypertension (PAH) at Weeks 28, 40, 52, 64, 76, 88, 100, 112 and 124
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, 100, 112 and 124
Population: Efficacy analysis set was used in this analysis. Here, 'Overall number of participants analyzed' specifies number of participants who completed Part 1 of the study and continued treatment with Sildenafil in Part 2 of the study and 'Number analyzed' = Participants evaluable for this outcome measure for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 3
Participants
  Baseline: Class I | 1
  Baseline: Class II | 2
  Baseline: Class III | 0
  Baseline: Class IV | 0
  Week 28: Improved | 1
  Week 28: No Change | 2
  Week 28: Worsened | 0
  Week 40: Improved | 1
  Week 40: No Change | 2
  Week 40: Worsened | 0
  Week 52: Improved | 1
  Week 52: No Change | 2
  Week 52: Worsened | 0
  Week 64: Improved: number analyzed (Participants) | 2
  Week 64: Improved | 1
  Week 64: No Change: number analyzed (Participants) | 2
  Week 64: No Change | 1
  Week 64: Worsened: number analyzed (Participants) | 2
  Week 64: Worsened | 0
  Week 76: Improved: number analyzed (Participants) | 2
  Week 76: Improved | 1
  Week 76: No Change: number analyzed (Participants) | 2
  Week 76: No Change | 0
  Week 76: Worsened: number analyzed (Participants) | 2
  Week 76: Worsened | 1
  Week 88: Improved: number analyzed (Participants) | 1
  Week 88: Improved | 1
  Week 88: No Change: number analyzed (Participants) | 1
  Week 88: No Change | 0
  Week 88: Worsened: number analyzed (Participants) | 1
  Week 88: Worsened | 0
  Week 100: Improved: number analyzed (Participants) | 1
  Week 100: Improved | 1
  Week 100: No Change: number analyzed (Participants) | 1
  Week 100: No Change | 0
  Week 100: Worsened: number analyzed (Participants) | 1
  Week 100: Worsened | 0
  Week 112: Improved: number analyzed (Participants) | 1
  Week 112: Improved | 1
  Week 112: No Change: number analyzed (Participants) | 1
  Week 112: No Change | 0
  Week 112: Worsened: number analyzed (Participants) | 1
  Week 112: Worsened | 0
  Week 124: Improved: number analyzed (Participants) | 1
  Week 124: Improved | 1
  Week 124: No Change: number analyzed (Participants) | 1
  Week 124: No Change | 0
  Week 124:Worsened: number analyzed (Participants) | 1
  Week 124:Worsened | 0

9. Secondary Outcome: Change From Baseline in Brain Natriuretic Peptide (BNP) at Week 52 and End of Treatment (EOT)
Description: BNP is produced by ventricular cardiomyocytes. It causes reduction in preload and blood pressure by vasodilatation.
Time Frame: Baseline, Week 52 and End of treatment (maximum duration of treatment: 119.6 weeks)
Population: Efficacy analysis set included all participants who received at least 1 dose of study drug.Here 'Overall number of participants analyzed' specifies number of participants who completed Part 1 of the study and continued treatment with Sildenafil in Part 2 of the study.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Sildenafil
Number analyzed (Participants) | 3
picograms per milliliter
  Baseline | 100.17 (151.478)
  Change at Week 52 | -85.17 (155.088)
  Change at EoT | -85.17 (155.088)

10. Secondary Outcome: Change From Baseline in N-terminal Pro Brain Natriuretic Peptide (NT Pro-BNP) at Week 52 and End of Treatment (EOT)
Description: as for outcome 7
Time Frame: Baseline, Week 52 and End of treatment (maximum duration of treatment: 119.6 weeks)
Population: EEfficacy analysis set included all participants who received at least 1 dose of study drug.Here 'Overall number of participants analyzed' specifies number of participants who completed Part 1 of the study and continued treatment with Sildenafil in Part 2 of the study.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Sildenafil
Number analyzed (Participants) | 3
picograms per milliliter
  Baseline | 841.73 (1323.533)
  Change at Week 52 | -754.90 (1335.370)
  Change at EoT | -754.90 (1335.370)

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline upto 28 days after last dose of study drug (maximum duration of treatment: 119.6 weeks)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
Participants
  AEs | 6
  SAEs | 0

12. Secondary Outcome: Number of Participants With Treatment-Emergent Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline upto 28 days after last dose of study drug (maximum duration of treatment: 119.6 weeks)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
Participants
  AEs | 3
  SAEs | 0

13. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure (BP) at Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, 100, 112 and 124
Description: BP measurement is recorded as supine and sitting systolic and diastolic systemic blood pressure: 1) Systolic blood pressure when heart is contracting and it is the maximum arterial pressure during contraction of left ventricle. 2) Diastolic BP when heart is relaxing and it is the minimum arterial pressure during relaxation and dilation of ventricles. Only those categories in which at least 1 participant had data were reported.
Time Frame: Baseline, Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, 100, 112 and 124
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, 'Number analyzed' = Participants evaluable for this outcome measure for specified categories.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
mmHg
  Baseline: Supine Systolic BP: number analyzed (Participants) | 5
  Baseline: Supine Systolic BP | 95.4 (13.41)
  Baseline: Supine Diastolic BP: number analyzed (Participants) | 5
  Baseline: Supine Diastolic BP | 55.8 (10.87)
  Baseline: Sitting Systolic BP: number analyzed (Participants) | 1
  Baseline: Sitting Systolic BP | 110.0
  Baseline: Sitting Diastolic BP: number analyzed (Participants) | 1
  Baseline: Sitting Diastolic BP | 60.0
  Change at Week 4: Supine Systolic BP: number analyzed (Participants) | 5
  Change at Week 4: Supine Systolic BP | 5.6 (9.91)
  Change at Week 4: Supine Diastolic BP: number analyzed (Participants) | 5
  Change at Week 4: Supine Diastolic BP | 1.6 (13.65)
  Change at Week 4: Sitting Systolic BP: number analyzed (Participants) | 1
  Change at Week 4: Sitting Systolic BP | 16.0
  Change at Week 4: Sitting Diastolic BP: number analyzed (Participants) | 1
  Change at Week 4: Sitting Diastolic BP | 23.0
  Change at Week 8: Supine Systolic BP: number analyzed (Participants) | 4
  Change at Week 8: Supine Systolic BP | 7.8 (14.93)
  Change at Week 8: Supine Diastolic BP: number analyzed (Participants) | 4
  Change at Week 8: Supine Diastolic BP | 2.3 (12.28)
  Change at Week 8: Sitting Systolic BP: number analyzed (Participants) | 1
  Change at Week 8: Sitting Systolic BP | -6.0
  Change at Week 8: Sitting Diastolic BP: number analyzed (Participants) | 1
  Change at Week 8: Sitting Diastolic BP | -3.0
  Change at Week 16: Supine Systolic BP: number analyzed (Participants) | 3
  Change at Week 16: Supine Systolic BP | 7.7 (17.62)
  Change at Week 16: Supine Diastolic BP: number analyzed (Participants) | 3
  Change at Week 16: Supine Diastolic BP | -1.3 (12.22)
  Change at Week 16: Sitting Systolic BP: number analyzed (Participants) | 1
  Change at Week 16: Sitting Systolic BP | 8.0
  Change at Week 16: Sitting Diastolic BP: number analyzed (Participants) | 1
  Change at Week 16: Sitting Diastolic BP | 10.0
  Change at Week 28: Supine Systolic BP: number analyzed (Participants) | 3
  Change at Week 28: Supine Systolic BP | 7.0 (19.31)
  Change at Week 28: Supine Diastolic BP: number analyzed (Participants) | 3
  Change at Week 28: Supine Diastolic BP | 1.7 (9.29)
  Change at Week 40: Supine Systolic BP: number analyzed (Participants) | 2
  Change at Week 40: Supine Systolic BP | -7.5 (3.54)
  Change at Week 40: Supine Diastolic BP: number analyzed (Participants) | 2
  Change at Week 40: Supine Diastolic BP | 2.0 (0.00)
  Change at Week 52: Supine Systolic BP: number analyzed (Participants) | 2
  Change at Week 52: Supine Systolic BP | 2.0 (15.56)
  Change at Week 52: Supine Diastolic BP: number analyzed (Participants) | 2
  Change at Week 52: Supine Diastolic BP | 10.0 (5.66)
  Change at Week 64: Supine Systolic BP: number analyzed (Participants) | 1
  Change at Week 64: Supine Systolic BP | 1.0
  Change at Week 64: Supine Diastolic BP: number analyzed (Participants) | 1
  Change at Week 64: Supine Diastolic BP | 8.0
  Change at Week 76: Supine Systolic BP: number analyzed (Participants) | 1
  Change at Week 76: Supine Systolic BP | -13.0
  Change at Week 76: Supine Diastolic BP: number analyzed (Participants) | 1
  Change at Week 76: Supine Diastolic BP | 3.0

14. Secondary Outcome: Change From Baseline in Heart Rate at Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, 100, 112 and 124
Description: Only those categories in which at least 1 participant had data were reported.
Time Frame: Baseline, Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, 100, 112 and 124
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
beats per minute (bpm)
  Baseline: Supine Heart rate: number analyzed (Participants) | 5
  Baseline: Supine Heart rate | 100.2 (15.91)
  Baseline: Sitting Heart rate: number analyzed (Participants) | 1
  Baseline: Sitting Heart rate | 96.0
  Change at Week 4: Supine Heart rate: number analyzed (Participants) | 5
  Change at Week 4: Supine Heart rate | -1.0 (12.08)
  Change at Week 4: Sitting Heart rate: number analyzed (Participants) | 1
  Change at Week 4: Sitting Heart rate | -22.0
  Change at Week 8: Supine Heart rate: number analyzed (Participants) | 4
  Change at Week 8: Supine Heart rate | -0.5 (9.11)
  Change at Week 8: Sitting Heart rate: number analyzed (Participants) | 1
  Change at Week 8: Sitting Heart rate | 0.0
  Change at Week 16: Supine Heart rate: number analyzed (Participants) | 3
  Change at Week 16: Supine Heart rate | 3.0 (28.69)
  Change at Week 16: Sitting Heart rate: number analyzed (Participants) | 1
  Change at Week 16: Sitting Heart rate | 4.0
  Change at Week 28: Supine Heart rate: number analyzed (Participants) | 3
  Change at Week 28: Supine Heart rate | 6.7 (14.36)
  Change at Week 40: Supine Heart rate: number analyzed (Participants) | 2
  Change at Week 40: Supine Heart rate | 10.0 (16.97)
  Change at Week 52: Supine Heart rate: number analyzed (Participants) | 2
  Change at Week 52: Supine Heart rate | -2.0 (11.31)
  Change at Week 64: Supine Heart rate: number analyzed (Participants) | 1
  Change at Week 64: Supine Heart rate | 17.0
  Change at Week 76: Supine Heart rate: number analyzed (Participants) | 1
  Change at Week 76: Supine Heart rate | -8.0

15. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory abnormality criteria: Hematology (hemoglobin, hematocrit, red blood cell count [less than {<}]0.8*lower limit of normal [LLN]; platelets <0.5*LLN, greater than [>]1.75*upper limit of normal [ULN], white blood cells <0.6*LLN, >1.5*ULN; lymphocytes, neutrophils <0.8*LLN, >1.2*ULN, eosinophils, basophils, monocytes >1.2*ULN); liver function (total and direct bilirubin >1.5*ULN, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase >3.0*ULN, total protein, albumin <0.8*LLN, >1.2*ULN); renal (creatinine, blood urea nitrogen >1.3*ULN); electrolytes (sodium <0.95*LLN, >1.05*ULN, potassium, chloride <0.9*LLN, >1.1*ULN; other (glucose <0.6*LLN or >1.5*ULN ); urinalysis (dipstick) urine glucose, urine protein, urine blood/Hemoglobin, [greater than or equal to {>=}1].
Time Frame: Baseline up-to End of treatment (maximum duration of treatment: 119.6 weeks)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
Participants | 4

16. Secondary Outcome: Number of Participants With Clinically Significant 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Criteria for clinically significant abnormality in ECG parameters: Maximum corrected QT interval (QTc) from 450 millisecond (msec) to less than (<) 480 msec, Maximum QTcB interval (Bazett's Correction) from 450 msec to <480 msec, Maximum QTcF interval (Fredericia's Correction) from 450 msec to <480 msec, maximum QTc interval increase from baseline of 30 msec to <60 msec and >=60 msec.
Time Frame: Screening, Week 16, Week 52 and End of treatment (maximum duration of treatment: 119.6 weeks)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
Participants
  Screening | 4
  Week 16 | 5
  Week 52: number analyzed (Participants) | 2
  Week 52 | 1
  End of Treatment: number analyzed (Participants) | 3
  End of Treatment | 1

17. Secondary Outcome: Number of Participants With Ocular Examination Abnormalities
Description: Ocular examination measures included external examination of the eye, funduscopy, assessments of visual acuity, and color vision. Ocular examination findings were considered abnormal based on investigator's decision.
Time Frame: Screening up to end of treatment (maximum duration of treatment: 119.6 weeks)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
Participants | 0

18. Secondary Outcome: Change From Baseline in Pulmonary Artery Systolic and Diastolic Pressure at Week 16
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
mmHg
  Baseline: Systolic Pressure | 82.5 (35.51)
  Baseline: Diastolic Pressure | 42.0 (18.19)
  Change at Week 16: Systolic Pressure: number analyzed (Participants) | 4
  Change at Week 16: Systolic Pressure | -9.8 (18.01)
  Change at Week 16: Diastolic Pressure: number analyzed (Participants) | 4
  Change at Week 16: Diastolic Pressure | -3.5 (13.99)

19. Secondary Outcome: Change From Baseline in Systemic Artery Systolic and Diastolic Pressure at Week 16
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
mmHg
  Baseline: Systolic Pressure | 95.3 (15.20)
  Baseline: Diastolic Pressure | 60.2 (19.30)
  Change at Week 16: Systolic Pressure: number analyzed (Participants) | 4
  Change at Week 16: Systolic Pressure | 0.3 (10.21)
  Change at Week 16: Diastolic Pressure: number analyzed (Participants) | 4
  Change at Week 16: Diastolic Pressure | -1.5 (14.25)

20. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) at Week 16
Description: The resistance to blood flow through the pulmonary circulation is known as PVR. It is largely influenced by the caliber of the pulmonary arteries and capillaries and was measured in terms of Wood units. Wood unit =80 dyne*seconds per centimetre^5 (dyne*sec/cm^5).
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Wood units
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
Wood units
  Baseline | 21.372 (11.3408)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | -6.145 (10.3499)

21. Secondary Outcome: Change From Baseline in Right Atrial Pressure (RAP) at Week 16
Description: RAP is the blood pressure in the right atrium of the heart. It reflects the amount of blood returning to the heart and the ability of the heart to pump the blood into the arterial system. RAP was measured using a pressure transducer positioned at the mid-axillary line with the participant in the supine position.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
mmHg
  Baseline | 6.5 (2.88)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | 1.3 (2.36)

22. Secondary Outcome: Change From Baseline in Pulmonary Capillary Wedge Pressure (PCWP) at Week 16
Description: PCWP was measured by pulmonary artery catheterization and provided an indirect measure of left atrial pressure.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
mmHg
  Baseline | 8.5 (0.84)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | 2.5 (1.00)

23. Secondary Outcome: Change From Baseline in Cardiac Output (CO) at Week 16
Description: Cardiac output is simply the amount of blood pumped by the heart per minute.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter per minute
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
liter per minute
  Baseline | 2.620 (0.9879)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | 0.420 (0.9076)

24. Secondary Outcome: Change From Baseline in Cardiac Index (CI) at Week 16
Description: Cardiac index is a hemodynamic parameter that relates the cardiac output from left ventricle in one minute to BSA, thus relating heart performance to the size of the individual. CI was calculated as cardiac output in systemic circulation divided by BSA.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter per minute per meter square
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
liter per minute per meter square
  Baseline | 3.070 (0.7460)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | 0.658 (1.8912)

25. Secondary Outcome: Change From Baseline in Systemic Vascular Resistance (SVR) at Week 16
Description: The resistance to blood flow through the systemic circulation is known as SVR. This can be used in measuring blood pressure, blood flow and cardiac function and measured in terms of Wood units. Wood unit =80 dyne*seconds per centimetre^5 (dyne*sec/cm^5).
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Wood units
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
Wood units
  Baseline | 26.545 (3.0768)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | -3.403 (4.4409)

26. Secondary Outcome: Change From Baseline in Systemic Vascular Resistance Index (SVRI) at Week 16
Description: SVRI equals systemic vascular resistance (SVR) times BSA. SVR is the resistance to blood flow through the systemic circulation and it was measured in Wood units. Wood unit =80 dyne*seconds per centimetre^5 (dyne*sec/cm^5).
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Wood units*meter^2
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
Wood units*meter^2
  Baseline | 23.855 (12.1480)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | -2.378 (3.9096)

27. Secondary Outcome: Change From Baseline in Mixed Venous Oxygen Saturation (SvO2) at Week 16
Description: SvO2 is the percentage of mixed venous oxygen (amount of oxygen bound to hemoglobin in venous blood). Change from baseline in percentage of mixed venous oxygen was reported in this outcome measure.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of mixed venous oxygen
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
percentage of mixed venous oxygen
  Baseline | 65.30 (8.549)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | 5.38 (12.426)

28. Secondary Outcome: Change From Baseline in Arterial Oxygen Saturation (SaO2) at Week 16
Description: SaO2 is the percentage of arterial oxygen (amount of oxygen bound to hemoglobin in arterial blood). Change from baseline in percentage of arterial oxygen was reported in this outcome measure.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of arterial oxygen
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
percentage of arterial oxygen
  Baseline | 95.08 (2.730)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | -0.80 (1.691)

29. Other Pre Specified Outcome: Maximum Observed Plasma Concentration (Cmax) of Sildenafil and UK-103,320
Description: UK-103,320 was the main metabolite of Sildenafil and was produced by cytochrome P450 3A4.
Time Frame: Pre-dose (0 hour) on Week 4, 8, 16 and 1, 2, 4, 8 hours post-dose on Week 16
Population: Pharmacokinetic (PK) parameter analysis set included all participants who have at least 1 of PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
nanogram per milliliter (ng/mL)
  Sildenafil | 138.1 (73)
  UK-103,320 | 73.66 (48)

30. Other Pre Specified Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Sildenafil and UK-103,320
Description: UK-103,320 was the main metabolite of Sildenafil and was produced by cytochrome P450 3A4.
Time Frame: Pre-dose (0 hour) on Week 4, 8, 16 and 1, 2, 4, 8 hours post-dose on Week 16
Population: PK parameter analysis set included all participants who have at least 1 of PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per millimeter
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
nanogram*hour per millimeter
  Sildenafil | 338.9 (54)
  UK-103,320 | 210.2 (74)

31. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Sildenafil and UK-103,320
Description: UK-103,320 was the main metabolite of Sildenafil and was produced by cytochrome P450 3A4.
Time Frame: Pre-dose (0 hour) on Week 4, 8, 16 and 1, 2, 4, 8 hours post-dose on Week 16
Population: PK parameter analysis set included all participants who have at least 1 of PK parameters of interest.
Measure: Median (Full Range); unit: hour
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
hour
  Sildenafil | 1.00 [1.00 to 1.97]
  UK-103,320 | 1.00 [1.00 to 1.97]

32. Other Pre Specified Outcome: Terminal Half Life (t1/2) of Sildenafil and UK-103,320
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half of its original concentration. UK-103,320 was a main metabolite of sildenafil and was produced by cytochrome P450 3A4.
Time Frame: Pre-dose (0 hour) on Week 4, 8, 16 and 1, 2, 4, 8 hours post-dose on Week 16
Population: PK parameter analysis set included all participants who have at least 1 of PK parameters of interest. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Median (Full Range); unit: hour
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
hour
  Sildenafil: number analyzed (Participants) | 2
  Sildenafil | 1.785 [1.63 to 1.94]
  UK-103,320: number analyzed (Participants) | 3
  UK-103,320 | 2.110 [2.04 to 3.26]

33. Other Pre Specified Outcome: Apparent Oral Clearance (CL/F) of Sildenafil
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Pre-dose (0 hour) on Week 4, 8, 16 and 1, 2, 4, 8 hours post-dose on Week 16
Population: PK parameter analysis set included all participants who have at least 1 of PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
liter per hour | 41.73 (77)

34. Other Pre Specified Outcome: Apparent Volume of Distribution (Vz/F) of Sildenafil
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Pre-dose (0 hour) on Week 4, 8, 16 and 1, 2, 4, 8 hours post-dose on Week 16
Population: PK parameter analysis set included all participants who have at least 1 of PK parameters of interest. Here, Overall Number of participants analyzed signifies those participants who were evaluable for this measure.
Measure: Median (Full Range); unit: liter
Arm/Group | Sildenafil
Number analyzed (Participants) | 2
liter | 77.90 [62.4 to 93.4]

35. Other Pre Specified Outcome: Change From Baseline in Ratio of Acceleration Time to Ejection Time (AcT/ET) at Week 16
Description: Acceleration time and ejection time are quantitative Doppler parameters and ratio of acceleration time to ejection time is a useful tool to evaluate the severity of aortic stenosis.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
ratio
  Baseline | 0.3038 (0.09675)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | 0.0175 (0.10261)

36. Other Pre Specified Outcome: Change From Baseline in Right Ventricular Tei Index at Week 16
Description: The right ventricular Tei Index is an index of myocardial performance. It is defined as the sum of isovolumic contraction time and isovolumic relaxation time divided by the ejection time.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
ratio
  Baseline: number analyzed (Participants) | 3
  Baseline | 0.7540 (0.48602)
  Change at Week 16: number analyzed (Participants) | 2
  Change at Week 16 | -0.0440 (0.37618)

37. Other Pre Specified Outcome: Change From Baseline in Right Ventricular Size at Week 16
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
centimeter (cm)
  Baseline | 3.37 (1.216)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | -0.40 (0.408)

38. Other Pre Specified Outcome: Change From Baseline in Tricuspid Valve Annulus Size at Week 16
Description: The tricuspid valve lies between the right atrium and the right ventricle and is placed in a more apical position than the mitral valve. The annulus separates the right atrium from the right ventricle. Change from baseline in tricuspid valve annulus size (in cm) was reported in this outcome measure.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
cm
  Baseline | 2.190 (0.5636)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | -0.103 (0.3727)

39. Other Pre Specified Outcome: Change From Baseline in Tricuspid Regurgitation - Pressure Gradient (TR-PG) Peak at Week 16
Description: Tricuspid regurgitation (insufficiency) is the failure of the tricuspid valve to close properly during systole, leading to the leaking of blood from the right ventricle into the right atrium. Change from baseline in TR-PG peak (in mmHg) was reported in this outcome measure.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
mmHg
  Baseline: number analyzed (Participants) | 5
  Baseline | 73.0 (39.31)
  Change at Week 16: number analyzed (Participants) | 2
  Change at Week 16 | -6.0 (33.94)

40. Other Pre Specified Outcome: Change From Baseline in Pulmonary Regurgitation - Pressure Gradient (PR-PG) End-Diastole at Week 16
Description: Pulmonary regurgitation (PR) or insufficiency is a valvular heart disease characterized by an incomplete closure of the pulmonary valve leading to a diastolic reflux into the right ventricle. Change from baseline in PR-PG end-diastole (in mmHg) was reported in this outcome measure.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
mmHg
  Baseline: number analyzed (Participants) | 3
  Baseline | 29.0 (14.73)
  Change at Week 16: number analyzed (Participants) | 2
  Change at Week 16 | 3.5 (13.44)

41. Other Pre Specified Outcome: Number of Participants With Pericardial Effusion
Description: Pericardial effusion is the presence of an abnormal amount of fluid in the pericardial cavity, as determined by echocardiography.
Time Frame: Baseline up to Week 16
Population: Efficacy analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
participants | 0

42. Other Pre Specified Outcome: Change From Baseline in Tricuspid Annular Plane Systolic Excursion (TAPSE) at Week 16
Description: Tricuspid annular plane systolic excursion is a parameter depicting global right ventricular function. Change from baseline in TAPSE (in cm) was reported in this outcome measure.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Sildenafil
Number analyzed (Participants) | 6
cm
  Baseline | 1.47 (0.437)
  Change at Week 16: number analyzed (Participants) | 4
  Change at Week 16 | 0.18 (0.320)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (maximum duration of treatment: 119.6 weeks)
Arm/Group | Sildenafil
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil (N=6)
Cardiac failure (Cardiac disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Feeling abnormal (General disorders) | 1
Bronchitis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 1
Ammonia increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Weight increased (Investigations) | 1
Headache (Nervous system disorders) | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 1 — As the event is gender specific, only female participants were evaluated.
Erection increased (Reproductive system and breast disorders) | 1 — As the event is gender specific, only female participants were evaluated.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Vision blurred (Eye disorders) | 1
Visual acuity reduced transiently (Eye disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Molluscum contagiosum (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Blood urine present (Investigations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.